CLINICAL TRIAL: NCT05085262
Title: Cardiovascular Disease and Outcomes Among Patients With SARS-CoV-2 (COVID-19) Infection During Hospital Admission and Post Discharge
Brief Title: Cardiovascular Disease and Outcomes Among Patients With SARS-CoV-2 Infection (COVID-19)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Dinesh Thavendiranathan, Cardiologist, University Health Network, Toronto
Other Study IDs: COVID-19 Study 20-5453
Record Dates: First submitted 2021-09-10; First posted 2021-10-20 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: COVID-19 Respiratory Infection
MeSH Terms: interventions — Echocardiography; Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples will be collected at time of admission to ER in those who are discharged after assessment and at three time points during admission in patients who are admitted for measurement of blood biomarkers
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Mild Disease: Those assessed as an outpatient or discharged from the emergency department and never admitted elsewhere based on patient history
  Interventions: Diagnostic Test: Bloodwork, Echocardiogram, PET/MRI
- Moderate Disease: Those admitted but never requiring transfer to ICU or similar advanced care setting
  Interventions: Diagnostic Test: Bloodwork, Echocardiogram, PET/MRI
- Severe Disease: Those requiring admission to ICU or other advanced care settings (i.e. other Level 2 beds)
  Interventions: Diagnostic Test: Bloodwork, Echocardiogram, PET/MRI
- Control Group: Those with a negative COVID-19 and no history of COVID-19
  Interventions: Diagnostic Test: Bloodwork, Echocardiogram, MRI

INTERVENTIONS:
Diagnostic Test: Bloodwork, Echocardiogram, PET/MRI — The study will use blood samples from COVID biobank at University Health Network. Samples will be collected at time of admission to ER in patients discharged after assessment and at three time points during admission in patients who are admitted for measurement of blood biomarkers. Echocardiography studies will be assessed for structural and functional abnormalities. All included patients will have prospective short-term follow-up (3-6 months) for assessment of clinical events and subclinical cardiovascular disease. 50 patients who had clinical cardiac MRI at our center within 5 years prior to COVID-19 (January 2015-January 2020) and have since tested positive for COVID-19 will be recruited for research cardiac MRI to compare changes between baseline (pre-COVID) and follow-up (post-COVID imaging). A subgroup of 50 patients will undergo cardiac PET/MRI at 1-3 months post COVID-19 diagnosis to evaluate for myocardial inflammation and other imaging markers of cardiac injury.
  Groups: Mild Disease; Moderate Disease; Severe Disease
Diagnostic Test: Bloodwork, Echocardiogram, MRI — The study will involve use of blood samples from the COVID biobank at UHN (University Health Network) for measurement of blood biomarkers. Echocardiography Studies will be systematically assessed for structural and functional abnormalities. All included patients assessment of clinical events and subclinical cardiovascular disease.
  Groups: Control Group

SUMMARY:
The coronavirus disease of 2019 (COVID-19) has affected over 2.4 million individuals worldwide and has resulted in >171,000 deaths. Cardiovascular disease (CVD) is an important contributor to death in these patients. Those who develop cardiac injury during infection have a 4-fold increased risk of death. Furthermore, pre-existing CVD or cardiovascular risk factors (e.g. diabetes, hypertension) are associated with worse outcomes. Given the recent emergence of this disease, there is limited understanding of:

(i) the risk factors for cardiovascular events, (ii) blood biomarkers for early recognition, and drug targeting, of patients at risk of adverse outcomes, and (iii) the short term subclinical and clinical cardiovascular manifestations in those who survive to discharge.

DETAILED DESCRIPTION:
COVID-19 and CVD: On March 11, 2020 the coronavirus disease of 2019 (COVID-19), which is caused by infection with SARS-CoV-2 virus, was declared a pandemic by the World Health Organization. Incredibly, >2,400,000 cases and >171,000 deaths have been reported globally as of April 21, 2020. While the overall case fatality is ~5%, the mortality rate is dramatically higher in selected populations, particularly in those with preexistent and/or new-onset cardiovascular disease (CVD)2. Early reports suggest that up to 20-28% of hospitalized patients with confirmed COVID-19 (COVID-19+) have evidence of cardiovascular injury, defined as troponin elevation with or without other cardiovascular manifestations such as ischemia, ventricular arrhythmias, and left ventricular dysfunction (LVD). While SARS-CoV-1 virus can directly infect the heart4, it is still not clear whether this is the case for SARS-CoV-2. Nevertheless, cardiovascular injury may result from indirect damage secondary to hypoxemia, sepsis, cytokine release, endothelial injury or from direct myocardial involvement. Regardless of the mechanism, early studies demonstrate that cardiovascular injury is associated with a 4-fold increased risk of death, independent of age, cardiovascular risk factors, preexistent CVD, non-CVD comorbidities, and ARDS (Acute Respiratory Distress Syndrome).The presence of CVD and cardiac injury appear to have a synergistic effect on adverse prognosis.5 However, the long-term consequences of this acute cardiovascular injury are not known, but are likely to be significant. Therefore, understanding early markers of cardiovascular injury, their association with adverse events (cardiovascular and non-cardiovascular) and post-discharge cardiovascular consequences of COVID-19 will allow better care of these patients.

Rationale for the study This study will address the above-mentioned knowledge gaps by focusing on patients with a broad spectrum of disease severity. It will include patients admitted to the hospital (sicker group) and those discharged from the emergency department (healthier group). It will focus on endothelial and cardiac blood biomarkers to facilitate early recognition of patients at risk for adverse events and characterize in-hospital and post-discharge cardiovascular sequelae of COVID-19. Ultimately, the intention is to identify patients at risk, reduce in-hospital and post-discharge adverse events, and determine the need for longer-term CVD prevention strategies and follow-up in survivors.

Endothelial cells (ECs) line every blood vessel within the human body and play a key role in CVD. During early COVID-19 infection ECs in the alveolar unit in the lung are likely injured due to the antiviral response of the lung cells. Furthermore, ECs also have receptors on their surface that can allow the virus to enter into the circulation and travel to other organs, including the heart. Therefore, damage to the endothelium, both directly or due to the body's antiviral inflammatory response, can contribute to cardiac injury and poor overall outcomes.

Cardiac injury can be identified by the release of cardiac markers in the blood such as troponin I and B-type natriuretic peptides, which can often be seen before overt heart dysfunction occurs. Therefore, we propose that measurement of both endothelial activation and cardiac-specific markers from patient's blood early after infection (i.e. at presentation) and during hospital admission, can serve as an indicator of early cardiovascular injury. Correlating these findings with abnormalities in cardiac functional tests as well as cardiovascular and non-cardiovascular adverse outcomes during admission and follow-up, will help us use these biomarkers to institute targeted prevention strategies.

Given that the majority of patients (>95%) who are infected with the virus survive, and cardiac injury during the infection is common, it is likely that there is significant unrecognized cardiac injury in survivors. This is often undetected during admission or in those discharged from the emergency department (ER) due to inability to perform complete cardiovascular assessment. To understand subclinical cardiovascular injury, all patients will be brought back 3-6 months for complete cardiac assessment using echocardiography, cardiac MRI, and bloodwork. This knowledge will enable strategies to prevent subsequent overt CVD events and to determine the need for further investigations and long-term follow-up in COVID-19 survivors.

ELIGIBILITY:
Inclusion Criteria:

1. COVID-19+ confirmed by RT-PCR (Reverse Transcriptase - Polymerase Chain Reaction).
2. Age ≥ 18 years.

Exclusion Criteria:

1. Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will enroll a total of 300 participants seen at UHN and SMH - 250 patients who have confirmed COVID-19 and 50 COVID-19- patients as a control group.
Sampling Method: Non-Probability Sample
Enrollment: 251 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Prevalence of abnormalities on cardiac MRI | 3 months
  The prevalence of myocardial inflammation and damage on cardiac MRI will be compared between patients with COVID-19 and controls.

SECONDARY OUTCOMES:
Prevalence of abnormalities on transthoracic echocardiography | 3 months
  The prevalence of cardiac abnormalities on echocardiography will be compared between patients with COVID-19 and controls.
Number of participants with abnormal blood biomarkers | 3 months
  Circulating blood markers of acute cardiac damage, endothelial and coagulation pathway activation, and microRNA biomarker profiles will be compared between patients admitted to the hospital versus those discharged from the emergency department
Major adverse cardiac and cerebrovascular events (MACCE) | 12 months
  MACCE is a composite of: Myocardial infarction; Unplanned coronary revascularization (PCI, CABG, thrombolysis) ; Heart failure hospitalization; Stroke (ischemic only); Arrhythmia requiring hospitalization; Cardiovascular death
Prevalence of myocardial inflammation on PET/MRI | 1 months
  The prevalence of myocardial inflammation on PET/MRI will be evaluated in a subgroup of 50 patients recovered from COVID-19.

CONTACTS AND LOCATIONS:
Overall Officials: Dinesh Thavendiranathan, Principal Investigator — University Health Network, Toronto; Kate Hanneman, Principal Investigator — University Health Network, Toronto; Kathryn Howe, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hospital, UHN, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided